CLINICAL TRIAL: NCT04363840
Title: The LEAD COVID-19 Trial: Low-risk, Early Aspirin and Vitamin D to Reduce COVID-19 Hospitalizations
Acronym: LEAD COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-063
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: COVID; Vitamin D Deficiency; Coagulopathy; Disseminated Intravascular Coagulation
MeSH Terms: conditions — Vitamin D Deficiency; Hemostatic Disorders; Disseminated Intravascular Coagulation | interventions — Aspirin; Vitamin D

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Observation (No Intervention)
- Aspirin 81 mg (Experimental)
  Interventions: Drug: Aspirin 81 mg
- Aspirin + vitamin D (Experimental): Offered to COVID-19 patients who are vitamin D deficient AND randomized to aspirin
  Interventions: Drug: Aspirin 81 mg; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Aspirin 81 mg — Aspirin 81 mg to be taken orally once daily for 14 days.
  Arms: Aspirin + vitamin D; Aspirin 81 mg
Dietary Supplement: Vitamin D — Vitamin D 50,000 IU to be taken orally once weekly for 2 weeks
  Arms: Aspirin + vitamin D

SUMMARY:
Although the novel SARS-CoV-2 virus (COVD-19) is classified as an acute respiratory infection, emerging data show that morbidity and mortality are driven by disseminated intravascular coagulopathy. Untreated CAC leads to microangiopathic thromboses, causing multiple systems organ failure and consuming enormous healthcare resources. Identifying strategies to prevent CAC are therefore crucial to reducing COVID-19 hospitalization rates.

The pathogenesis of CAC is unknown, but there are major overlaps between severe COVID-19 and vitamin D insufficiency (VDI). We hypothesize that VDI is a major underlying contributor to CAC. Preliminary data from severe COVID-19 patients in New Orleans support this hypothesis. The purpose of the proposed multi-center, prospective, randomized controlled trial is to test the hypothesis that low-risk, early treatment with aspirin and vitamin D in COVID-19 can mitigate the prothrombotic state and reduce hospitalization rates.

DETAILED DESCRIPTION:
Although the novel SARS-CoV-2 virus (COVD-19) is classified as an acute respiratory infection, emerging data show that morbidity and mortality are driven by disseminated intravascular coagulopathy. Data from Wuhan showed that COVID-19-associated coagulopathy (CAC) was present in 71% of deaths vs. 0.4% of survivors. Untreated CAC leads to microangiopathic thromboses, causing multiple systems organ failure and consuming enormous healthcare resources. Identifying strategies to prevent CAC are therefore crucial to reducing COVID-19 hospitalization rates.

The high prevalence of CAC in severely ill COVID-19 patients led the American Society of Hematology to recommend that all hospitalized COVID-19 patients be prophylactically anticoagulated. However, there are no data and no recommendations regarding outpatient prevention of CAC.

The pathogenesis of CAC is unknown. Given the demographic, geographic, pathologic, and treatment overlap between severe COVID-19 and vitamin D insufficiency (VDI), we hypothesize that VDI is a major underlying contributor to CAC. Preliminary data from critically ill COVID-19 patients in New Orleans support this hypothesis. Furthermore, mouse models of VDI developed aggravated multiorgan thrombus formation after lipopolysaccharide injection; this phenotype parallels CAC.

Given these lines of evidence, the purpose of the proposed multi-center, prospective, randomized controlled trial is to test the hypothesis that low-risk, early treatment with aspirin and vitamin D in COVID-19 (The LEAD COVID-19 Trial) can mitigate the prothrombotic state and reduce hospitalization rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Written informed consent
* New (within 24 hours) COVID-19 diagnosis

Exclusion Criteria:

* Pregnant patients or Prisoners
* History of GI bleeding or peptic ulcer disease, or spontaneous bleeding from other sites; History of thrombocytopenia; History of chronic kidney disease; Concurrent use of nonsteroidal anti-inflammatory drugs, or steroids.
* Hypervitaminosis D and associated risk factors: Renal failure, Liver failure, Hyperparathyroidism, Sarcoidosis, Histoplasmosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | 2 weeks
  Hospitalization for COVID-19 symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Frank H Lau, MD, Principal Investigator — LSUHSC-NO

REFERENCES:
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818